CLINICAL TRIAL: NCT03615534
Title: Efficacy and Safety of Extended Release Niacin-Fenofibrate Combination and Monotherapy for the Treatment of Atherogenic Dyslipidemia in Obese Females
Brief Title: Extended Release Niacin and Fenofibrate for the Treatment of Atherogenic Dyslipidemia in Obese Females
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lewai Sharki Abdulaziz, MSc PhD (Other)
Collaborators: Al-Kindy College of Medicine (Other)
Responsible Party: Sponsor-Investigator, Lewai Sharki Abdulaziz, MSc PhD, Assistant Professor, Al-Kindy College of Medicine
Organization: Al-Kindy College of Medicine (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 1 Al-KindyCM
Record Dates: First submitted 2018-07-27; First posted 2018-08-06 (Actual); Results first posted 2018-10-12 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Atherogenic Dyslipidemia; Obesity Associated Disorder
Keywords: Extended Release Niacin; Fenofibrate; treatment; Obesity; Atherogenic Dyslipidemia
MeSH Terms: conditions — Obesity | interventions — Fenofibrate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Placebo (Placebo Comparator): Non-responders to four-week therapeutic lifestyle changes run-in period, will start to receive an after lunch daily single placebo capsule for eight weeks.
  Interventions: Other: Therapeutic Lifestyle Changes; Other: Placebo
- Fenofibrate Monotherapy (Active Comparator): Non-responders to four-week therapeutic lifestyle changes run-in period, will start to receive an after lunch 200mg daily single dose of fenofibrate (Lipanthyl® 200 mg micronized fenofibrate capsule, Abbott Laboratories Fournier) for eight weeks.
  Interventions: Other: Therapeutic Lifestyle Changes; Drug: Fenofibrate
- WMER Niacin Monotherapy (Active Comparator): Non-responders to four-week therapeutic lifestyle changes run-in period, will start to receive a night-time 500 mg daily single dose of Wax Matrix Extended Release Niacin (WMER Niacin, ENDUR-ACIN®500mg, Endurance Products Company, Oregon USA) for one week, titrated up to 1000 mg by adding a daily morning-time ENDUR-ACIN®500mg tablet for the next seven weeks.
  Interventions: Other: Therapeutic Lifestyle Changes; Dietary Supplement: Wax Matrix Extended Release Niacin (WMER Niacin)
- Combination Therapy (Active Comparator): Non-responders to four-week therapeutic lifestyle changes run-in period, will start to receive an after lunch 200mg daily single dose of fenofibrate for eight weeks, in combination with a night-time 500 mg daily single dose of WMER Niacin for one week, titrated up to 1000mg by adding a daily morning-time ENDUR-ACIN®500mg tablet for the next seven weeks.
  Interventions: Other: Therapeutic Lifestyle Changes; Drug: Fenofibrate; Dietary Supplement: Wax Matrix Extended Release Niacin (WMER Niacin)

INTERVENTIONS:
Other: Therapeutic Lifestyle Changes — Four-week therapeutic lifestyle changes run-in period, comprising individualized moderate physical activity and total calories reduction.
Other: Placebo
  Arms: Placebo
Drug: Fenofibrate
  Other Names: Lipanthyl
  Arms: Combination Therapy; Fenofibrate Monotherapy
Dietary Supplement: Wax Matrix Extended Release Niacin (WMER Niacin)
  Other Names: ENDUR-ACIN®
  Arms: Combination Therapy; WMER Niacin Monotherapy

SUMMARY:
Atherogenic Dyslipidemia (AD) is a risk-conferring lipid/lipoprotein profile that comprises a higher proportion of small LDL particles, reduced HDL-C, and increased triglycerides. It is characteristically seen in patients with obesity, metabolic syndrome, insulin resistance, and type 2 diabetes mellitus and has emerged as an important marker for the increased cardiovascular disease (CVD) risk observed in these populations.

Optimal cardiovascular risk reduction in patients exhibiting the lipid triad of AD requires integrated pharmacotherapy to normalize HDL-C, Triglyceride (TG) and LDL-C levels. Recent studies have focused on optimizing treatment for AD and compare the efficacy and tolerability of combined lipid-altering drug based therapies, however, an optimal pharmacologic approach has not yet been established.

The present study was intended to evaluate the restorative efficacy of Extended Release Niacin (ER Niacin) and Fenofibrate as mono and combination therapies , as well as their safety and tolerability in females with obesity-induced AD.

DETAILED DESCRIPTION:
Study Setting:

The present study is a single blinded placebo-controlled randomized clinical trial, in which target individuals were obese females (BMI≥30 kg/m2), within the age of 20-60 years, attending the Obesity research and therapy unit of Al-Kindy College of Medicine, University of Baghdad (Baghdad, Iraq), throughout the period from 1st October 2014 to 15th March 2015.

Study Protocol:

Target individuals with fulfill devoid of exclusion criteria, were further screened and only candidates with conventional diagnosis of AD, as confirmed by a fasting serum TG >150 mg/dl coincide with an HDL-C of less than 50 mg/dl, were considered to be enrolled. Finally, and successive to a comprehensible concise for the expected benefits and side effects on top of the commitment to the entire protocol, eligible candidates settled for participation were provided with a written informed consent.

Enrollment:

1. Therapeutic Lifestyle Changes (TLC) Run-in Period: Each and every eligible candidate was enrolled in a four-week TLC run-in (or lead-in) period to exclude responders and to obtain baseline data for non-responders prior to randomization.
2. Randomization and Treatment Allocation: TLC non-responders with persistent AD were randomly allocated to one of the four treatment arms. In order to ensure a periodical balance among all study groups in the course of treatment allocation, permuted-block randomization with a block size of four was implemented and the system produced by this approach was adopted for the sequential random assignment of patients to treatment arms. .

Discontinuation of Treatment:

Although the absence of published consensus on drug discontinuation in the face of laboratory abnormalities has permitted a spectrum of indefinite decisions, mainly driven by clinical experience, clinical status and tolerability of the patient. For the present study discontinuation of treatment is considered if:

1. Adverse events including flushing, nausea, vomiting, muscle pain, or dizziness turn sever enough to surpass patient's tolerability.
2. Estimated glomerular filtration rate (eGFR) is reduced to ˂ 60ml/min per 1.73 m2 indicating renal insufficiency.
3. Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) increased to>3 Upper Limit of Normal (ULN) with the appearance of nausea, vomiting, fatigue, right upper quadrant pain or tenderness, fever, and/or rash.
4. Serum uric acid exceeds the critical value of 6mg/dl.

Assessment of Treatments Responses:

Responses to the different treatments arms, in terms of efficacy and safety, are assessed by analyzing clinical and laboratory data collected at each visit over the entire course of the study, including a thorough medical history and previous medication records.

Statistical Analysis:

All statistical analyses were executed via the statistical package SPSS version 17.0 (SPSS, Inc.). Prior to analysis, Shapiro-Wilk test was used for assessing the normality of distributions for continuous variables, with the data expressed as the mean ± standard error (SE). Analysis of variance (ANOVA) was applied to compare the means of baseline characteristics among different treatments groups. Comprising the influence of the baseline level as a covariate, analysis of covariance (ANCOVA), embracing the least significant difference (LSD) for pair-wise comparison, was applied to assess treatment effects and safety profiles among different arms. Results were evaluated in terms of adjusted end line levels and percent changes from baseline levels. Multivariate Analysis of Covariance (MANCOVA), on the other hand, with further adjustments for relevant covariates was conducted whenever needed. Probability of less than 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* BMI≥30 kg/m2.
* Conventional diagnosis of atherogenic dyslipidemia, confirmed by a fasting serum TG more than150 mg/dl coincide with an HDL-C of less than 50 mg/dl.

Exclusion Criteria:

* The use of any antilipidemic medication.
* Findings suggestive for renal dysfunction (eGFR˂60ml/min per 1.73 m2).
* Findings suggestive for hepatic insufficiency (ALT and/or AST˃2ULN).
* Clinical or laboratory findings suggestive for thyroid dysfunction.
* Established diagnosis of Diabetes Mellitus.
* History of gout, hyperuricemia, or on hypouricemic agents.
* Active peptic ulcer.
* Pregnancy, or nursing mothers.
* Alcohol or tobacco consumption.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 161 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lewai S Abdulaziz, MSc PhD, Study Chair — Al-Kindy college of Medicine, University of Baghdad; May S Al-Sabbagh, MSc, Study Chair — College of Pharmacy, University of Baghdad; Marwah S Attar, MSc, Study Director — College of Pharmacy, University of Baghdad; Faris A Khazaal, FRCP, Principal Investigator — Al-Kindy college of Medicine, University of Baghdad
Locations (2):
- Iraq (2):
  - Al Kindy College of Medicine, University of Baghdad, Baghdad
  - Lewai S Abdulaziz, Baghdad

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (table, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months and ending 24 months following article publication
Access Criteria: Anyone who wishes to access the data, to achieve aims in the approved proposal or for meta-analysis. The data will be available in our college's data warehouse up to 24 months following article publication.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Obese females (BMI≥30 kg/m2), within the age of 20-60 years, attending the Obesity research and therapy unit of Al-Kindy College of Medicine, Baghdad, Iraq, throughout the period from 1st October 2014 to 15th March 2015, were screened for preliminary eligibility.
Pre-assignment Details: Out of the 161 obese females settled for participation, Atherogenic dyslipidemia (AD) was diagnosed in 69(42.9%) patients, all of whom were enrolled in Therapeutic Lifestyle Changes (TLC) run-in period. AD was averted by TLC in 12(17.4%) patients. The remaining 57(82.6%) non-responding patients were randomly allocated to one of the four study arms.
Groups:
- Placebo: Non-responders to four-week therapeutic lifestyle changes run-in period, will start to receive an after lunch daily single placebo capsule for eight weeks.
  Therapeutic Lifestyle Changes: Four-week therapeutic lifestyle changes run-in period, comprising individualized moderate physical activity and total calories reduction.
  Placebo
- Fenofibrate Monotherapy: Non-responders to four-week therapeutic lifestyle changes run-in period, will start to receive an after lunch 200mg daily single dose of fenofibrate (Lipanthyl® 200 mg micronized fenofibrate capsule, Abbott Laboratories Fournier) for eight weeks.
  Therapeutic Lifestyle Changes: Four-week therapeutic lifestyle changes run-in period, comprising individualized moderate physical activity and total calories reduction.
  Fenofibrate
- WMER Niacin Monotherapy: Non-responders to four-week therapeutic lifestyle changes run-in period, will start to receive a night-time 500 mg daily single dose of Wax Matrix Extended Release Niacin (WMER Niacin, ENDUR-ACIN®500mg, Endurance Products Company, Oregon USA) for one week, titrated up to 1000 mg by adding a daily morning-time ENDUR-ACIN®500mg tablet for the next seven weeks.
  Therapeutic Lifestyle Changes: Four-week therapeutic lifestyle changes run-in period, comprising individualized moderate physical activity and total calories reduction.
  Wax Matrix Extended Release Niacin (WMER Niacin)
- Combination Therapy: Non-responders to four-week therapeutic lifestyle changes run-in period, will start to receive an after lunch 200mg daily single dose of fenofibrate for eight weeks, in combination with a night-time 500 mg daily single dose of WMER Niacin for one week, titrated up to 1000mg by adding a daily morning-time ENDUR-ACIN®500mg tablet for the next seven weeks.
  Therapeutic Lifestyle Changes: Four-week therapeutic lifestyle changes run-in period, comprising individualized moderate physical activity and total calories reduction.
  Fenofibrate
  Wax Matrix Extended Release Niacin (WMER Niacin)
Period: Overall Study
Arm/Group | Placebo | Fenofibrate Monotherapy | WMER Niacin Monotherapy | Combination Therapy
Started | 14 | 15 | 14 | 14
Completed | 12 | 15 | 14 | 13
Not Completed | 2 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Fenofibrate Monotherapy | WMER Niacin Monotherapy | Combination Therapy | Total
Number analyzed (Participants) | 12 | 15 | 14 | 13 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (2.5) | 37.3 (2.0) | 36.6 (2.1) | 40.2 (2.2) | 37.6 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 14 | 13 | 54
  Male | 0 | 0 | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Weight (in Kilograms) and Height (in Meters) were measured using a portable stadiometer with movable head piece typically mounted on balanced beam scale (Segma, Germany). Body mass index (BMI) is the relative weight for height and it was calculated according to formula bellow:
  BMI=Weight (Kg) / Height2 (m)
  kg/m^2 | 38.9 (2.1) | 41.5 (1.7) | 42.0 (1.7) | 39.7 (1.8) | 40.6 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: Changes Serum Triglyceride Levels
Description: Assessments involve the measurement of serum Triglyceride (TG) level.
Time Frame: Treatments effects were assessed by two events, baseline investigations conducted before randomization and end line investigations at the end of the eighth week of treatments.
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Placebo | Fenofibrate Monotherapy | WMER Niacin Monotherapy | Combination Therapy
Number analyzed (Participants) | 12 | 15 | 14 | 13
mg/dl
  Baseline TG levels | 223.1 (23.4) | 241.2 (19.1) | 227.0 (19.7) | 267.2 (20.5)
  Adjusted End line TG levels | 220.2 (12.8) | 133.7 (11.4) | 164.0 (11.4) | 136.1 (12.0)
Statistical Analysis 1: Comparison: Placebo vs Fenofibrate Monotherapy vs WMER Niacin Monotherapy vs Combination Therapy; Multivariate Analysis of Covariance (MANCOVA), was applied to assess treatment effects among different arms, comprising the influence of the baseline TG level as a covariate, with further adjustments for baseline HDL-C, ApoA1levels; Test type: Superiority; p = 0.0001, MANCOVA — Results were evaluated in terms of adjusted end line TG levels, embracing the least significant difference (LSD) for pair-wise comparison. Probability of less than 0.05 was considered statistically significant; Covariates appearing in MANCOVA model are evaluated at the following baseline values: TG= 240.4 mg/dl, HDL-C = 31.8 mg/dl, ApoA1 = 144.6 mg/dl

2. Primary Outcome: Changes in Serum Lipoprotein Cholesterol Levels
Description: Assessments involve the measurement of serum Total (TC), High density lipoprotein (HDL-C) and direct Low density lipoprotein (d-LDL-C) cholesterol levels.
  Serum non HDL-C levels is calculated by subtracting HDL-C from TC. Serum Remnant cholesterol (RC) is calculated by subtracting HDL-C and d-LDL-C from TC.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Placebo | Fenofibrate Monotherapy | WMER Niacin Monotherapy | Combination Therapy
Number analyzed (Participants) | 12 | 15 | 14 | 13
mg/dl
  Baseline TC | 203.1 (11.4) | 190.7 (9.3) | 189.1 (9.6) | 219.5 (10.0)
  Baseline HDL-C | 30.9 (2.1) | 32.1 (1.7) | 34.2 (1.8) | 29.7 (1.8)
  Baseline d-LDL-C | 120.0 (7.5) | 108.9 (6.2) | 120.1 (6.4) | 129.3 (6.6)
  Baseline non HDL-C | 172.3 (11.3) | 158.6 (9.2) | 154.9 (9.5) | 189.7 (9.9)
  Baseline RC | 52.3 (8.4) | 49.7 (6.8) | 34.9 (7.1) | 60.5 (7.3)
  Adjusted End line TC | 198.4 (7.4) | 171.1 (6.7) | 177.3 (6.6) | 179.9 (6.4)
  Adjusted End line HDL-C | 32.0 (1.4) | 37.2 (1.3) | 38.3 (1.3) | 42.8 (1.3)
  Adjusted End line d-LDL-C | 115.7 (6.6) | 103.6 (5.9) | 103.3 (5.9) | 115.0 (6.2)
  Adjusted End line non HDL-C | 166.4 (7.7) | 134.1 (6.9) | 138.7 (6.9) | 136.3 (7.2)
  Adjusted End line RC | 50.7 (4.8) | 30.3 (4.3) | 35.7 (4.3) | 22.1 (4.5)
Statistical Analysis 1: Comparison: Placebo vs Fenofibrate Monotherapy vs WMER Niacin Monotherapy vs Combination Therapy; Multivariate Analysis of Covariance (MANCOVA), was applied to assess treatment effects among different arms, comprising the influence of the baseline TC level as a covariate, with further adjustments for baseline Non HDL-C and d-LDL-C; Test type: Superiority; p = 0.060, MANCOVA — Results were evaluated in terms of adjusted end line TC levels, embracing the least significant difference (LSD) for pair-wise comparison. Probability of less than 0.05 was considered statistically significant; Covariates appearing in MANCOVA model are evaluated at the following baseline values: TC=199.9 mg/dl, Non HDL-C= 168.0 mg/dl, d-LDL-C= 119.1 mg/dl
Statistical Analysis 2: Comparison: Placebo vs Fenofibrate Monotherapy vs WMER Niacin Monotherapy vs Combination Therapy; Multivariate Analysis of Covariance (MANCOVA), was applied to assess treatment effects among different arms, comprising the influence of the baseline HDL-C level as a covariate, with further adjustments for baselineTG, ApoA1levels; Test type: Superiority; p = 0.0001, MANCOVA — Results were evaluated in terms of adjusted end line HDL-C levels, embracing the least significant difference (LSD) for pair-wise comparison. Probability of less than 0.05 was considered statistically significant; Covariates appearing in MANCOVA model are evaluated at the following baseline values: HDL-C = 31.8 mg/dL,TG= 240.4 mg/dL, ApoA1 = 144.6 mg/dL
Statistical Analysis 3: Comparison: Placebo vs Fenofibrate Monotherapy vs WMER Niacin Monotherapy vs Combination Therapy; Multivariate Analysis of Covariance (MANCOVA), was applied to assess treatment effects among different arms, comprising the influence of the baseline d-LDL-C level as a covariate, with further adjustments for baseline TC and Non HDL-C; Test type: Superiority; p = 0.334, MANCOVA — Results were evaluated in terms of adjusted end line d-LDL-C levels, embracing the least significant difference (LSD) for pair-wise comparison. Probability of less than 0.05 was considered statistically significant; Covariates appearing in MANCOVA model are evaluated at the following baseline values: d-LDL-C= 119.1 mg/dl.TC=199.9 mg/dl, Non HDL-C= 168.0 mg/dl,
Statistical Analysis 4: Comparison: Placebo vs Fenofibrate Monotherapy vs WMER Niacin Monotherapy vs Combination Therapy; Multivariate Analysis of Covariance (MANCOVA), was applied to assess treatment effects among different arms, comprising the influence of the baseline Non HDL-C level as a covariate, with further adjustments for baseline TC and d-LDL-C; Test type: Superiority; p = 0.012, MANCOVA — Results were evaluated in terms of adjusted end line Non HDL-C levels, embracing the least significant difference (LSD) for pair-wise comparison. Probability of less than 0.05 was considered statistically significant; Covariates appearing in MANCOVA model are evaluated at the following baseline values: Non HDL-C= 168.0 mg/dl,TC=199.9 mg/dl, d-LDL-C= 119.1 mg/dl
Statistical Analysis 5: Comparison: Placebo vs Fenofibrate Monotherapy vs WMER Niacin Monotherapy vs Combination Therapy; Multivariate Analysis of Covariance (MANCOVA), was applied to assess treatment effects among different arms, comprising the influence of the baseline RC level as a covariate, with further adjustments for baselineTC, Non HDL-C, d-LDL-C, and ApoB; Test type: Superiority; p = 0.001, MANCOVA — Results were evaluated in terms of adjusted end line RC levels, embracing the least significant difference (LSD) for pair-wise comparison. Probability of less than 0.05 was considered statistically significant; Covariates appearing in MANCOVA model are evaluated at the following baseline values:RC=48.9,TC=199.9, Non HDL-C=168.0, d-LDL-C=119.1, ApoB=133.1mg/dl

3. Primary Outcome: Changes in Serum Apolipoprotein Levels
Description: Assessments involve the measurement of serum Apolipoprotein A1 (Apo A1) and B (Apo B) levels.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Placebo | Fenofibrate Monotherapy | WMER Niacin Monotherapy | Combination Therapy
Number analyzed (Participants) | 12 | 15 | 14 | 13
mg/dl
  Baseline Apo A1 | 130.8 (8.7) | 143.8 (7.1) | 150.1 (7.4) | 150.0 (7.7)
  Baseline Apo B | 134.1 (7.5) | 141.8 (6.1) | 123.0 (6.3) | 133.1 (6.6)
  Adjusted End line Apo A1 | 130.2 (10.4) | 155.9 (9.3) | 134.2 (9.3) | 162.3 (9.7)
  Adjusted End line Apo B | 124.7 (6.4) | 106.7 (5.7) | 111.1 (5.7) | 101.7 (6.0)
Statistical Analysis 1: Comparison: Placebo vs Fenofibrate Monotherapy vs WMER Niacin Monotherapy vs Combination Therapy; Multivariate Analysis of Covariance (MANCOVA), was applied to assess treatment effects among different arms, comprising the influence of the baseline ApoA1 level as a covariate, with further adjustments for baseline TG and HDL-C levels; Test type: Superiority; p = 0.058, MANCOVA — Results were evaluated in terms of adjusted end line ApoA1 levels, embracing the least significant difference (LSD) for pair-wise comparison. Probability of less than 0.05 was considered statistically significant; Covariates appearing in MANCOVA model are evaluated at the following baseline values: ApoA1 = 144.6 mg/dl, TG= 240.4 mg/dl, HDL-C = 31.8 mg/dl
Statistical Analysis 2: Comparison: Placebo vs Fenofibrate Monotherapy vs WMER Niacin Monotherapy vs Combination Therapy; Multivariate Analysis of Covariance (MANCOVA), was applied to assess treatment effects among different arms, comprising the influence of the baseline ApoB level as a covariate, with further adjustments for baselineTC, Non HDL-C, dLDL-C, and RC; Test type: Superiority; p = 0.067, MANCOVA — Results were evaluated in terms of adjusted end line ApoB levels, embracing the least significant difference (LSD) for pair-wise comparison. Probability of less than 0.05 was considered statistically significant; Covariates appearing in MANCOVA model are evaluated at the following baseline values:ApoB=133.1, RC=48.9,TC=199.9, Non HDL-C=168.0, d-LDL-C=119.1mg/dl

4. Secondary Outcome: Changes in Serum Fasting Glucose Levels.
Description: Assessments involve the measurement of serum fasting glucose levels.
Time Frame: Changes from baseline were assessed at the end eighth week of treatments.
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Placebo | Fenofibrate Monotherapy | WMER Niacin Monotherapy | Combination Therapy
Number analyzed (Participants) | 12 | 15 | 14 | 13
mg/dl
  Baseline serum fasting glucose | 93.5 (3.9) | 98.9 (3.2) | 94.6 (3.3) | 94.7 (3.4)
  Adjusted End line serum fasting glucose | 91.3 (2.3) | 91.7 (2.0) | 100.1 (2.1) | 87.3 (2.1)
Statistical Analysis 1: Comparison: Placebo vs Fenofibrate Monotherapy vs WMER Niacin Monotherapy vs Combination Therapy; Analysis of Covariance (ANCOVA), was applied to assess treatment effects among different arms, comprising the influence of the baseline FSG level as a covariate; Test type: Superiority; p = 0.001, ANCOVA — Results were evaluated in terms of adjusted end line FSG levels, embracing the least significant difference (LSD) for pair-wise comparison. Probability of less than 0.05 was considered statistically significant; Covariates appearing in ANCOVA model are evaluated at the following baseline values: FSG= 95.7 mg/dl

5. Secondary Outcome: Changes in Estimated Glomerular Filtration Rate (eGFR)
Description: Assessments involve the measurement of serum creatinine which is used to calculate eGFR using the CKD-EPI equation (2009) .
Time Frame: Changes from baseline were assessed at the end of the eighth week of treatments.
Measure: Mean (Standard Error); unit: ml/min per 1.73 m^2
Arm/Group | Placebo | Fenofibrate Monotherapy | WMER Niacin Monotherapy | Combination Therapy
Number analyzed (Participants) | 12 | 15 | 14 | 13
ml/min per 1.73 m^2
  Baseline eGFR | 89.8 (4.8) | 86.5 (3.9) | 91.0 (4.1) | 85.2 (4.2)
  Adjusted End line eGFR | 83.1 (3.4) | 83.2 (3.1) | 82.9 (3.2) | 79.2 (3.3)
Statistical Analysis 1: Comparison: Placebo vs Fenofibrate Monotherapy vs WMER Niacin Monotherapy vs Combination Therapy; Analysis of Covariance (ANCOVA), was applied to assess treatment effects among different arms, comprising the influence of the baseline eGFR level as a covariate; Test type: Superiority; p = 0.786, ANCOVA — Results were evaluated in terms of adjusted end line eGFR levels, embracing the least significant difference (LSD) for pair-wise comparison. Probability of less than 0.05 was considered statistically significant; Covariates appearing in ANCOVA model are evaluated at the following baseline values: eGFR= 88.0 ml/min per 1.73 m^2

6. Secondary Outcome: Changes in Serum Uric Acid Levels
Description: Assessments involve the measurement of serum uric acid levels
Time Frame: Changes from baseline were assessed at the end of the eighth week of treatments.
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Placebo | Fenofibrate Monotherapy | WMER Niacin Monotherapy | Combination Therapy
Number analyzed (Participants) | 12 | 15 | 14 | 13
mg/dl
  Baseline serum uric acid | 4.45 (0.30) | 5.21 (0.24) | 4.87 (0.25) | 5.28 (0.26)
  Adjusted End line serum uric acid | 4.80 (0.25) | 4.0 (0.22) | 5.6 (0.23) | 3.9 (0.24)
Statistical Analysis 1: Comparison: Placebo vs Fenofibrate Monotherapy vs WMER Niacin Monotherapy vs Combination Therapy; Analysis of Covariance (ANCOVA), was applied to assess treatment effects among different arms, comprising the influence of the baseline serum uric acid level as a covariate; Test type: Superiority; p = 0.0001, ANCOVA — Results were evaluated in terms of adjusted end line serum uric acid levels, embracing the least significant difference (LSD) for pair-wise comparison. Probability of less than 0.05 was considered statistically significant; Covariates appearing in ANCOVA model are evaluated at the following baseline values: serum uric acid= 5.0 mg/dl

7. Secondary Outcome: Changes in Serum Enzymes Levels
Description: Assessments involve the measurement of serum enzymes including Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) and Creatine Kinase (CK) levels.
Time Frame: Changes from baseline were assessed at the end of the eighth week of treatments.
Measure: Mean (Standard Error); unit: IU/L
Arm/Group | Placebo | Fenofibrate Monotherapy | WMER Niacin Monotherapy | Combination Therapy
Number analyzed (Participants) | 12 | 15 | 14 | 13
IU/L
  Baseline AST | 17.1 (1.6) | 18.8 (1.3) | 17.0 (1.4) | 18.9 (1.4)
  Baseline ALT | 13.1 (1.4) | 16.3 (1.2) | 16.0 (1.2) | 17.8 (1.2)
  Baseline CK | 28.0 (4.7) | 29.1 (3.8) | 26.9 (4.0) | 28.0 (4.1)
  Adjusted End line AST | 18.9 (0.8) | 17.3 (0.8) | 18.0 (0.8) | 19.6 (0.8)
  Adjusted End line ALT | 15.4 (0.6) | 14.4 (0.5) | 16.4 (0.5) | 16.2 (0.6)
  Adjusted End line CK | 27.3 (4.7) | 34.9 (4.2) | 27.4 (4.4) | 28.2 (4.5)
Statistical Analysis 1: Comparison: Placebo vs Fenofibrate Monotherapy vs WMER Niacin Monotherapy vs Combination Therapy; Analysis of Covariance (ANCOVA), was applied to assess treatment effects among different arms, comprising the influence of the baseline AST level as a covariate; Test type: Other; p = 0.201, ANCOVA — Results were evaluated in terms of adjusted end line AST levels, embracing the least significant difference (LSD) for pair-wise comparison. Probability of less than 0.05 was considered statistically significant; Covariates appearing in ANCOVA model are evaluated at the following baseline values: AST= 18.1 IU/L
Statistical Analysis 2: Comparison: Placebo vs Fenofibrate Monotherapy vs WMER Niacin Monotherapy vs Combination Therapy; Analysis of Covariance (ANCOVA), was applied to assess treatment effects among different arms, comprising the influence of the baseline ALT level as a covariate; Test type: Superiority; p = 0.033, ANCOVA — Results were evaluated in terms of adjusted end line ALT levels, embracing the least significant difference (LSD) for pair-wise comparison. Probability of less than 0.05 was considered statistically significant; Covariates appearing in ANCOVA model are evaluated at the following baseline values: ALT= 16.0 IU/L
Statistical Analysis 3: Comparison: Placebo vs Fenofibrate Monotherapy vs WMER Niacin Monotherapy vs Combination Therapy; Analysis of Covariance (ANCOVA), was applied to assess treatment effects among different arms, comprising the influence of the baseline CK level as a covariate; Test type: Superiority; p = 0.511, ANCOVA — Results were evaluated in terms of adjusted end line CK levels, embracing the least significant difference (LSD) for pair-wise comparison. Probability of less than 0.05 was considered statistically significant; Covariates appearing in ANCOVA model are evaluated at the following baseline values: CK= 28.0 IU/L

8. Secondary Outcome: Changes in Systolic and Diastolic Blood Pressure
Description: Assessments involve the measurement of systolic and diastolic blood pressure. Patients were allowed to rest for 15 minutes in sitting position, and Walgreens Homedics WGNBPA-540 upper arm blood pressure monitor (Walgreens, China), was used for the measurement of blood pressure. Three consecutive readings were taken at 1 minute interval, and systolic and diastolic blood pressure were calculated as the mean of the last two readings.
Time Frame: Changes from baseline were assessed at the end of the eighth week of treatments.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Fenofibrate Monotherapy | WMER Niacin Monotherapy | Combination Therapy
Number analyzed (Participants) | 12 | 15 | 14 | 13
mmHg
  Baseline diastolic blood pressure | 80.7 (2.6) | 83.5 (2.1) | 76.1 (2.3) | 77.3 (2.4)
  Baseline systolic blood pressure | 120.7 (3.9) | 125.4 (3.1) | 118.5 (3.4) | 119.5 (3.5)
  Adjusted End line diastolic blood pressure | 79.5 (1.0) | 78.6 (0.9) | 80.3 (1.1) | 80.9 (1.1)
  Adjusted End line systolic blood pressure | 118.3 (2.1) | 117.4 (1.8) | 117.8 (2.2) | 118.8 (2.2)
Statistical Analysis 1: Comparison: Placebo vs Fenofibrate Monotherapy vs WMER Niacin Monotherapy vs Combination Therapy; Analysis of Covariance (ANCOVA), was applied to assess treatment effects among different arms, comprising the influence of the baseline diastolic blood pressure level as a covariate; Test type: Other; p = 0.434, ANCOVA — Results were evaluated in terms of adjusted end line diastolic blood pressure levels, embracing the least significant difference (LSD) for pair-wise comparison. Probability of less than 0.05 was considered statistically significant; Covariates appearing in ANCOVA model are evaluated at the following baseline values: diastolic blood pressure= 80.0 mmHg
Statistical Analysis 2: Comparison: Placebo vs Fenofibrate Monotherapy vs WMER Niacin Monotherapy vs Combination Therapy; Analysis of Covariance (ANCOVA), was applied to assess treatment effects among different arms, comprising the influence of the baseline systolic blood pressure level as a covariate; Test type: Superiority; p = 0.966, ANCOVA — Results were evaluated in terms of adjusted end line systolic blood pressure levels, embracing the least significant difference (LSD) for pair-wise comparison. Probability of less than 0.05 was considered statistically significant; Covariates appearing in ANCOVA model are evaluated at the following baseline values: systolic blood pressure= 121.5 mmHg

9. Secondary Outcome: Adverse Events
Description: Assessments comprise the total number of participants complicating and reporting muscle pain,flushing, nausea, vomiting, and dizziness.
  As part of the complete safety profile of each arm,other specific reported adverse event are presented in the Adverse Event Module.
Time Frame: Changes from baseline were assessed at the end of the eighth week of treatments.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fenofibrate Monotherapy | WMER Niacin Monotherapy | Combination Therapy
Number analyzed (Participants) | 12 | 15 | 14 | 13
Participants
  Muscle Pain | 0 | 0 | 0 | 1
  Flushing | 0 | 0 | 1 | 0
  Nausea/Vomiting | 0 | 0 | 3 | 1
  Dizziness | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to the end of the eighth week of treatments.
Arm/Group | Placebo | Fenofibrate Monotherapy | WMER Niacin Monotherapy | Combination Therapy
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/15 | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/15 | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 0/12 | 0/15 | 7/14 | 3/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | Fenofibrate Monotherapy (N=15) | WMER Niacin Monotherapy (N=14) | Combination Therapy (N=13)
Muscle Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Flushing (General disorders) | 0 | 0 | 1 | 0
Nausea/Vomiting (Gastrointestinal disorders) | 0 | 0 | 3 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
eGFR˂ 60ml/min per 1.73 m^2 (Renal and urinary disorders) | 0 | 0 | 0 | 0
ALT or AST >3ULN (Hepatobiliary disorders) | 0 | 0 | 0 | 0
Uric acid > 6 mg/dl (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No